CLINICAL TRIAL: NCT03448965
Title: Glycemic Disorders in Low Birth Weight Babies
Brief Title: Hypoglycemic and Hyperglycemic Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, martinamamdouh fahem, principle investigator, Assiut University
Other Study IDs: NGD
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Hypoglycemia in Newborn Infants; Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: random blood sugar — do random blood sugar at 0 hour - 2 hours- 4 hours and after 6 hours

SUMMARY:
Definition of low birth weight:

Low birth weight infants are those born weighing less than 2500 g. These are further subdivided into:

* Very Low Birth Weight : Birth weight <1,500 g
* Extremely Low Birth Weight : Birth weight <1,000 g Their survival is directly related to birth weight, with approximately 20% of those between 500 and 600 g and>90% of those between 1,250 and 1,500 g surviving. Perinatalcare has improved the rate of survival of low birth weight infants.

DETAILED DESCRIPTION:
Causes of low birth weight:

* Premature birth
* Intrauterine growth restriction, which are most often Due to different placental problems and health problems of the mother or new-born

RISK FACTORS:

* Age: Teen mothers have a much higher risk of having VLBW infant.
* Multiple birth babies are at increased risk of being VLBW because they often are premature. More than 50% of twins and other multiple gestations are VLBW if <15 years
* Maternal health: Women exposed to drugs, alcohol, and cigarettes during pregnancy are more likely to have low birth weight babies. Mothers of lower socioeconomic
* Race: African-American babies are twice as likely as Caucasian to be very low birth weight

ELIGIBILITY:
Inclusion Criteria:

* All neonates admitted to neonatology unit

  1. From 0-28 days
  2. Weighting less than 2500gm

Exclusion Criteria:

* Any neonate weighting more than 2500 gm

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all low birth weight babies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
glycemic disorders in low birth weight | one year
  to detect the prevelance of hypoglycemia and hyperglycemia in low birth weight babies by random blood sugar test

REFERENCES:
- [Background] Abdulkadir I, Hassan L, Abdullahi F, Sobowale AM, Akeredolu FD, Purdue S, Okpe M, Adewumi OA, Abdullahi U, Onadiran MA, Ogala WN. Outcome of Extremely Low Birth Weight Babies in Zaria; A Ten-Year Review. West Afr J Med. 2015 Jan-Mar;34(1):50-4. PMID 26902817
- [Background] Hays SP, Smith EO, Sunehag AL. Hyperglycemia is a risk factor for early death and morbidity in extremely low birth-weight infants. Pediatrics. 2006 Nov;118(5):1811-8. doi: 10.1542/peds.2006-0628. PMID 17079549
- [Background] Rozance PJ, Hay WW Jr. New approaches to management of neonatal hypoglycemia. Matern Health Neonatol Perinatol. 2016 May 10;2:3. doi: 10.1186/s40748-016-0031-z. eCollection 2016. PMID 27168942
- [Background] Eichenwald EC, Stark AR. Management and outcomes of very low birth weight. N Engl J Med. 2008 Apr 17;358(16):1700-11. doi: 10.1056/NEJMra0707601. No abstract available. PMID 18420502